CLINICAL TRIAL: NCT02191280
Title: The Ability of Antistax® to Improve Chronic Venous Insufficiency (CVI) I and II in Male and Female Patients: a Dose Response Study
Brief Title: Antistax® in Patients With Chronic Venous Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1138.2
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Antistax

ARMS (3):
- Antistax®, low dose (Experimental)
  Interventions: Drug: Antistax®, low dose
- Antistax®, high dose (Experimental)
  Interventions: Drug: Antistax®, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Antistax®, low dose
  Arms: Antistax®, low dose
Drug: Antistax®, high dose
  Arms: Antistax®, high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine the efficacy and tolerability of two dose levels of Antistax relative to placebo in patients suffering from CVI grade I or incipient grade II

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Between 25 and 75 years of age
* CVI I or CVI II (without expanded trophic disturbances)
* Willing and able to give written informed consent prior to participation in the study

Exclusion Criteria:

Concomitant disease(s) exclusion criteria:

* Decompensated cardiac insufficiency
* Edema not due to venous disease of the legs (e.g. latent cardiac insufficiency, renal insufficiency, lymph edema, etc)
* Peripheral arterial disease (ankle/arm pressure index < 0.9)
* Current acute phlebitis or thrombosis
* Renal insufficiency (Serum creatinine > 1.5 mg/dl)
* Liver disease (SGPT (ALAT) > 3x upper limit of normal)
* Other diseases: insulin-dependent diabetes mellitus, neuropathies, hyper- or hypocalcaemia, malignancies
* Anamnestic indications of diabetic microangiopathy or polyneuropathy
* Drug and/or alcohol abuse
* Severe climacteric complaints
* Immobility
* Avalvulia
* Klippel-Trénaunay-Weber-Syndrome (Naevus varicosis osteohypertrophicus, Haemangiectasia hypertrophicans)
* State after pulmonary embolism
* Recognized hypersensitivity to the trial drug ingredients
* Current florid venous ulcus
* Clinical indication for a necessary, specific phlebologic acute treatment, e.g. compressive treatment, phlebectomy, etc.

Previous treatment(s) exclusion criteria:

* Treatment with venous drugs within the last 4 weeks
* Treatment with laxatives which affect fluid or electrolyte balance within the last 8 days
* Changes in or unstable response to treatment with theophylline, diuretics, cardiac glycosides, ACE inhibitors or calcium antagonists within the last 8 days
* Changes in post-menopausal Hormone replacement within the last 2 months

Concomitant treatment/non-drug therapy exclusion criteria:

* Other venous drugs apart from the trial medication
* Compression therapy
* Venous surgery at the leg(s)
* Extensive use (on more than a total of 6 days during the entire trial) of laxatives which affect fluid or electrolyte balance
* Major surgery requiring full anesthesia

Other exclusion criteria:

* Previously studied under this protocol
* Participation in another clinical trial within the previous 90 days or during the present study
* Patients who have visited a sauna or had other thermal applications in the previous day before any visit
* Pregnant or nursing women or inadequate birth control methods (this applies to females of childbearing potential only)
* Patients considered as mentally ill as well as unable to work or with limited working ability, or unable (or only partially able) to follow the spoken or written explanations concerning the trial
* Patients in a bad general health state according to the investigator's judgment

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1998-04; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of limb volume | Baseline, day 84
  determined by water displacement

SECONDARY OUTCOMES:
Changes of limb volume | Baseline, days 42 and 98
  determined by water displacement
Measurement of calf circumference | Baseline, days 42, 84 and 98
  in centimeters
Measurement of ankle circumference | Baseline, days 42, 84 and 98
  in centimeters
Assessment of subjective symptoms on a visual analogue scale (VAS) | Baseline, days 42, 84 and 98
Assessment of global efficacy by patient on a 4-point verbal rating scale | days 42, 84 and 98
Assessment of global efficacy by investigator on a 4-point verbal rating scale | days 42, 84 and 98
Assessment of global tolerability by patient on a 4-point verbal rating scale | days 42, 84 and 98
Assessment of global tolerability by investigator on a 4-point verbal rating scale | days 42, 84 and 98
Number of patients with adverse events | up to 14 weeks

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449